CLINICAL TRIAL: NCT01194700
Title: Comparative Study of Lung Bioavailability of HFA-Seretide Via Current Spacer Devices in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAI008; 2007-003627-20 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: lung bioavailability; asthma; seretide; Spacer
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Evohaler (Experimental)
  Interventions: Drug: Seretide 250(8puffs) via Evohaler actuator; Drug: Seretide 250 (8 puffs)/placebo via Volumatic spacer; Drug: Seretide 250/placebo 8 puffs via Aerochamber Plus spacer; Drug: Seretide 250/placebo via Synchro-Breathe
- Volumatic spacer (Experimental)
  Interventions: Drug: Seretide 250(8puffs) via Evohaler actuator; Drug: Seretide 250 (8 puffs)/placebo via Volumatic spacer; Drug: Seretide 250/placebo 8 puffs via Aerochamber Plus spacer; Drug: Seretide 250/placebo via Synchro-Breathe
- Aerochamber Plus (Experimental)
  Interventions: Drug: Seretide 250(8puffs) via Evohaler actuator; Drug: Seretide 250 (8 puffs)/placebo via Volumatic spacer; Drug: Seretide 250/placebo 8 puffs via Aerochamber Plus spacer; Drug: Seretide 250/placebo via Synchro-Breathe
- Synchro-Breathe (Experimental)
  Interventions: Drug: Seretide 250(8puffs) via Evohaler actuator; Drug: Seretide 250 (8 puffs)/placebo via Volumatic spacer; Drug: Seretide 250/placebo 8 puffs via Aerochamber Plus spacer; Drug: Seretide 250/placebo via Synchro-Breathe

INTERVENTIONS:
Drug: Seretide 250(8puffs) via Evohaler actuator — 8 puffs of Seretide250/Placebo via Evohaler actuator
  Other Names: Advair
Drug: Seretide 250 (8 puffs)/placebo via Volumatic spacer — 8 puffs of Seretide 250/placebo via volumatic spacer
  Other Names: Advair
Drug: Seretide 250/placebo 8 puffs via Aerochamber Plus spacer — Seretide 250/placebo 8 puffs via Aerochamber Plus
  Other Names: Advair
Drug: Seretide 250/placebo via Synchro-Breathe — Seretide 250/placebo 8puffs via breath actuated Synchro-Breathe device
  Other Names: Advair

SUMMARY:
The purpose of this study is to determine the effect of plastic spacers and breath actuated spacers on respirable drug delivery of combination steroid inhaler (Seretide/Advair) and whether electrostatic charge within plastic spacers has a clinically relevant impact on the inhaled steroid delivery.

DETAILED DESCRIPTION:
Conventional plastic spacers are bulky and can be influenced by electrostatic charge, which can reduce respirable dose delivery especially when used brand new "out of the box". Breath actuated integrated vortex spacer (Synchro-Breathe) is a compact palm sized antistatic device with a vortex chamber which is designed to be more patient friendly and free from the effects of electrostatic charge. The systemic bioavailability from the lung of inhaled fluticasone and salmeterol is dependent on respirable dose delivery, and hence the performance of inhaler devices can be quantified by measuring the degree of adrenal suppression and fall in serum potassium(K) as surrogates for delivered lung dose. This study attempts to compares the systemic bioavailability from the lung in real life conditions for Fluticasone/Salmeterol combination (measured in terms of relative adrenal suppression and fall in serum K) via the breath actuated Synchro-Breathe device, pMDI( Seretide Evohaler), and Aerochamber Plus & Volumatic spacer used brand new "out of the box" in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers
2. Male or female 18-65
3. Informed Consent
4. Ability to comply with the requirements of the protocol

Exclusion Criteria:

1. No respiratory disease
2. Smokers
3. Recent respiratory tract infection (2 months).
4. Any other clinically significant medical condition such as unstable angina, acute myocardial infarction in the preceding 3 months, recent TIA/ CVA,that may endanger the health or safety of the participant, or jeopardise the protocol.
5. Any significant abnormal laboratory result as deemed by the investigators
6. Pregnancy, planned pregnancy or lactation
7. Known or suspected contra-indication to any of the IMP's
8. Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overnight Urinary Cortisol creatinine ratio | within 24 hours after study drug inhalation
  This outcome measure evaluates the amount of cortisol being suppressed after inhaled steroid administration. This helps to assess the systemic effect of steroid inhalation and therefore the propensity for adrenal suppression which is a noted adverse effect with high dose inhaled steroids

SECONDARY OUTCOMES:
Serum Potassium | 60 minutes post treatment
  The serum potassium is monitored 60 minutes post study drug inhalation to assess the systemic beta-2-adrenoreceptor metabolic response. Long acting beta agonists like Salmeterol exhibit dose related reduction in serum potassium.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Nair, Principal Investigator — University of Dundee; Brian J Lipworth, Study Director — University of Dundee
Locations (1):
- Asthma & Allergy Research Group, Department of cardiovascular & lung biology, Division of medicine, Ninewells Hospital & Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Result] Nair A, McKinlay L, Williamson P, Short P, Burns P, Lipworth BJ. Comparative lung bioavailability of fluticasone/salmeterol via a breath-actuated spacer and conventional plastic spacers. Eur J Clin Pharmacol. 2011 Apr;67(4):355-363. doi: 10.1007/s00228-010-0989-9. Epub 2011 Jan 15. PMID 21240480